CLINICAL TRIAL: NCT02038335
Title: HIV-Target Cell Response in Women Initiating Various Contraceptive Methods in High HIV-Incidence Areas: Zim CHIC
Acronym: Zim CHIC
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Zimbabwe (Other)
Responsible Party: Principal Investigator, Sharon Achilles, Principal Investigator and Protocol Chair, University of Pittsburgh
Other Study IDs: PRO13080550
Record Dates: First submitted 2014-01-08; First posted 2014-01-16 (Estimated); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Contraception; HIV; Immune Cells (Mucosal and Systemic); Microbiota
Keywords: immune cells; contraception; intrauterine device; IUD; copper; microbiota; DMPA; etonogestrel; subdermal implant; NET-EN; Jadelle; Implanon; Cyclofem
MeSH Terms: interventions — N,N-dimethyl-4-anisidine; norethindrone enanthate; Medroxyprogesterone Acetate; estradiol 17 beta-cypionate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, plasma archive, vaginal swabs, serum, cervicovaginal lavage fluid
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- DMPA: Depot medroxyprogesterone acetate
  Interventions: Drug: DMPA
- NET-EN: Norethisterone enantate
  Interventions: Drug: NET-EN
- MPA/E2: Medroxyprogesterone acetate and estradiol cypionate
  Interventions: Drug: MPA/E2
- LNG-I: Levonorgestrel subdermal implant
  Interventions: Device: LNG-I
- ENG-I: Etonogestrel subdermal implant
  Interventions: Device: ENG-I
- Cu-IUD: Copper IUD
  Interventions: Device: Cu-IUD

INTERVENTIONS:
Drug: DMPA — Depot medroxyprogesterone acetate
  Other Names: Depot medroxyprogesterone acetate (DMPA)
  Groups: DMPA
Drug: NET-EN — Norethisterone enantate
  Other Names: Norethisterone enantate (NET-EN)
  Groups: NET-EN
Drug: MPA/E2 — Medroxyprogesterone acetate and estradiol cypionate
  Other Names: Medroxyprogesterone acetate and estradiol cypionate (MPA/E2)
  Groups: MPA/E2
Device: LNG-I — Levonorgestrel subdermal implant
  Other Names: Levonorgestrel subdermal implant (LNG-I)
  Groups: LNG-I
Device: ENG-I — Etonogestrel subdermal implant
  Other Names: Etonogestrel subdermal implant (ENG-I)
  Groups: ENG-I
Device: Cu-IUD — Copper IUD
  Other Names: Copper IUD (Cu-IUD)
  Groups: Cu-IUD

SUMMARY:
This study is being done to understand if using birth control causes changes in the immune cells within the reproductive tract of healthy women. Immune cells are important because they help prevent infections from starting and help fight infections that have started. Immune cells are also the type of cells that HIV (human immunodeficiency virus) infects so understanding more about them will help to better understand how to prevent the spread of HIV.

Immune cells will be studied from the reproductive tract of women who want to start using one of the following contraceptives: Depo-Provera (DMPA), NET-EN, MPA/E2 (Cyclofem®), the levonorgestrel subdermal implant (Jadelle® ), the etonogestrel subdermal implant (Implanon® or Nexplanon® ) and the copper IUD.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 through 34 years (inclusive) at screening
* Non-pregnant women in general good health as determined by the site clinician
* Premenopausal with history of regular menstrual cycles (regular cycles defined as occurring every 21-35 days when not using hormones and with a variation of typical cycle length of no more than 5 days)
* Able and willing to provide written informed consent to be screened for and to take part in the study. Including willingness to undergo all study-related assessments and follow all study-related procedures
* Able and willing to provide adequate locator information
* HIV-uninfected based on testing performed by study staff at screening
* At screening and enrollment, agrees not to participate in other research studies involving drugs, medical devices, or vaginal products while enrolled in this trial

Exclusion Criteria:

* Use of any hormonal or intrauterine contraceptive method within 30 days of enrollment
* Use of DMPA or NET-EN within 10 months of enrollment
* Pregnancy or breastfeeding within 60 days of enrollment
* Surgical procedure involving the pelvis in the 30 days prior to enrollment (includes dilation and curettage, cryosurgery and biopsy of the vagina, vulva, cervix, and endometrium)
* Internal vaginal use of any device (includes sex toys, cervical caps, diaphragms, menstrual collection devices, and pessaries; excludes tampons and condoms) or product (includes N9, microbicide, douche, antifungal, steroid, or hormone) in the 30 days prior to enrollment
* New sexual partner within 90 days of enrollment
* Urogenital infection or suspected infection within 30 days of enrollment including:

symptomatic candidiasis, trichomoniasis, and symptomatic BV; or cervical infection, including N. gonorrhoeae, Chlamydia trachomatis, or mucopurulent cervicitis; syphilis; HSV lesions, or other sores (Note: seropositive HSV without active lesions will not be excluded); acute pelvic inflammatory disease; urinary tract infection; recent exposure to a partner with GC, CT, Trichomonas, syphilis, or NGU. Women who have had diagnosed genital infections should have completed treatment at least 30 days before the time of enrollment.

* Any history of immunosuppression (includes diabetes, HIV infection, and chronic steroid use)
* Antibiotic or antifungal therapy (vaginal or systemic) within 30 days of enrollment
* Menses or other vaginal bleeding at the time of Enrollment* (*Women who have vaginal bleeding at the scheduled Enrollment Visit may return at a different date to be re-examined and possibly enrolled provided they are still within the 90-day screening window and meet all criteria).
* Vaginal or anal intercourse within 2 days (48 hours) prior to enrollment
* Heterosexual intercourse since last menses that places the participant at risk of pregnancy (without condom use or sterilization of at least one partner)
* History of hysterectomy
* History of malignancy within the pelvis (includes uterus, cervix, vagina, and vulva)
* Contraindication, allergy or intolerance to use of the contraceptive desired by the participant
* Any condition that, in the opinion of the Investigator, would preclude provision of consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Healthy women, age 18-34 years, who are HIV negative and non-pregnant.
Sampling Method: Non-Probability Sample
Enrollment: 451 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Genital tract CD4 cells (number and % expressing CCR5) | Change from baseline at 3 months
  To quantify and characterize immune cell populations and HIV-tropic receptor expression in the genital tract and blood at baseline and after 1, 3 and 6 months of typical contraceptive use. Immune cell populations will be quantified and characterized using flow cytometry.

SECONDARY OUTCOMES:
Vaginal microbiota (key microbes) | Change from baseline at 3 months
  To describe the microflora of the genital tracts of healthy asymptomatic women before and after 1, 3 and 6 months of typical contraceptive use and to assess changes in the vaginal ecology within the first 6-months of contraceptive use. qPCR for key microflora and Nugent scores will be used.
Serum hemoglobin | Change from baseline at 6 months
  To objectively assess blood count before and at 1,3,and 6 months following initiation of each contraceptive method. Standard clinical complete blood count (CBC) will be obtained at each visit.
Serum concentration of estradiol and progesterone/progestin | Change from baseline at 3 months
  To assess relative serum concentrations of endogenous and exogenous sex hormones before and after contraceptive use. Hormonal concentrations will be assessed by measuring blood levels of estrogen and progesterone as well as blood levels of the contraceptive progestin corresponding to the cohort group for that participant.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Achilles, MD, PhD, Study Chair — University of Pittsburgh; Felix Mhlanga, MD, Principal Investigator — University of Zimbabwe, University of California San Francisco
Locations (1):
- UZ UCSF, Harare, Zimbabwe

REFERENCES:
- [Derived] Achilles SL, Meyn LA, Mhlanga FG, Matubu AT, Stoner KA, Beamer MA, Chirenje ZM, Hillier SL. Zim CHIC: A cohort study of immune changes in the female genital tract associated with initiation and use of contraceptives. Am J Reprod Immunol. 2020 Sep;84(3):e13287. doi: 10.1111/aji.13287. Epub 2020 Jun 25. PMID 32533883